CLINICAL TRIAL: NCT07205107
Title: Satisfaction, Adherence, Effectiveness, and Safety of Clindamycin Phosphate, Adapalene, and Benzoyl Peroxide Treatment in Patients With Acne Vulgaris: A Canadian Prospective Phase IV Study (CHARM)
Brief Title: Clindamycin Phosphate, Adapalene, and Benzoyl Peroxide Triple Combination Gel in Canadian Patients With Acne Vulgaris
Acronym: CHARM
Status: Recruiting | Type: Observational
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BHC-CAN-DERM-004
Record Dates: First submitted 2025-09-24; First posted 2025-10-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate; Adapalene; Benzoyl Peroxide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: clindamycin phosphate, adapalene and benzoyl peroxide — Topical treatment
  Other Names: CABTREO; IDP-126; Clindamycin Phosphate (1.2% w/w), Adapalene (0.15% w/w) and Benzoyl Peroxide (3.1% w/w)

SUMMARY:
The goal of this observational study is to learn about the effects of a treatment that contains clindamycin phosphate, adapalene, and benzoyl peroxide in people with acne. The main questions the study aims to answer are:

* How satisfied are people with this treatment?
* How well do people follow the treatment plan?
* How effective and safe is the treatment?
* How does the treatment affect quality of life?
* How do people use other skin care products, such as cleansers, moisturizers, and sunscreen, while using this treatment?

About 200 people aged 12 and older with acne across Canada will use the treatment as part of their regular care and answer questions about their experience over 20 weeks.

DETAILED DESCRIPTION:
This is a Phase IV, observational, prospective, multi-center study designed to evaluate treatment satisfaction, adherence, effectiveness, safety, tolerability, quality of life, and skin care product utilization patterns in patients with acne vulgaris who are treated with a topical gel containing clindamycin phosphate 1.2%, adapalene 0.15%, and benzoyl peroxide 3.1% in routine clinical practice across Canada. Approximately 200 patients aged 12 years and older will be enrolled at about 20 dermatology centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 12 years or older (unless minors are not permitted as per local regulations) who have been prescribed clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel as per the product monograph as part of routine clinical care for acne vulgaris but have not yet initiated treatment. The decision to prescribe clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel must be made prior to and independent of study participation.
* Patients and legally authorized representatives who are willing to provide written informed consent using an Institutional Review Board (IRB) or Independent Ethics Committee (IEC)-approved Informed Consent Form (ICF) in English or French. Patients who are less than the age of consent must sign an assent for the study and a parent, or a legal guardian must sign the informed consent.
* Patients who can read, understand, and communicate in English or French.

Patients must also meet the following additional inclusion criterion at the time of clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel initiation in order to be eligible for enrolment in the study:

* Patients have completed IRB or IEC-approved baseline ePROs (DermSat-7 and HUI2) after providing consent and prior to receiving their first dose of clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel.
* Patients have initiated clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel within 5 days of signed informed consent/assent.

Exclusion Criteria:

* Patients who have a contraindication to clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel as per the product monograph:

  1. Patients who are hypersensitive to clindamycin phosphate, to adapalene, to benzoyl peroxide or to any ingredient in the formulation or component of the container,
  2. Patients with a history of regional enteritis (Crohn's disease), ulcerative colitis, or antibiotic-associated colitis, and/or
  3. Pregnant women and women planning a pregnancy.
* Patients who, at the time of informed consent, are clear or almost clear (Investigator Global Assessment [IGA] = 0 or 1) or are on current acne therapy (topical or systemic, etc.)), or undergoing procedures (e.g., laser, photodynamic therapy) that could impact study results, as per the investigator's judgement.
* Patients who have any other serious and/or uncontrolled medical condition, and/or are receiving any medical therapy, that prohibits the patient from participating as per the investigator's judgement.
* Patients who have whey protein-triggered acne, drug-induced acne, occupational acne, acne associated with hidradenitis suppurativa or synovitis, acne, pustulosis, hyperostosis, and osteitis (SAPHO) syndrome, or acne related to hyperandrogenic states including polycystic ovary syndrome (PCOS).
* Patients who have conditions that mimic acne, including rosacea, folliculitis, perioral dermatitis, demodicosis.
* Patients who are not willing or able to complete electronic patient reported outcomes (ePROs) using an electronic device.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Canadian routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Treatment Satisfaction at Week-12 as assessed by DermSat-7 | Week 12
  To describe treatment satisfaction of clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel at Week-12 in patients with acne vulgaris in Canadian routine clinical practice, using mean DermSat-7 domain scores. The DermSat-7 is a dermatology-specific, 7-item questionnaire used to assess patient satisfaction with treatment across three domains: effectiveness, convenience, and overall satisfaction. Domain scores are transformed to a linear 0-100 scale, with higher scores indicating greater satisfaction.

SECONDARY OUTCOMES:
Treatment Satisfaction at Week-4, Week-8 and Week-20 as assessed by DermSat-7 | Week 4, Week 8 and Week 20
  To describe treatment satisfaction of clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel at Week-4, Week-8 and Week-20 in patients with acne vulgaris in Canadian routine clinical practice, using mean DermSat-7 domain scores. The DermSat-7 is a dermatology-specific, 7-item questionnaire used to assess patient satisfaction with treatment across three domains: effectiveness, convenience, and overall satisfaction. Domain scores are transformed to a linear 0-100 scale, with higher scores indicating greater satisfaction.
Change from Baseline in Treatment Satisfaction at Week-12 as assessed by DermSat-7 | Baseline and Week-12
  To describe change in treatment satisfaction at Week-12 following clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel initiation in patients with acne vulgaris in Canadian routine clinical practice, using mean DermSat-7 domain scores. The DermSat-7 is a dermatology-specific, 7-item questionnaire used to assess patient satisfaction with treatment across three domains: effectiveness, convenience, and overall satisfaction. Domain scores are transformed to a linear 0-100 scale, with higher scores indicating greater satisfaction.
Treatment Adherence at Week-4, Week-8, Week-12, and Week-20 | From Baseline to Week-20
  To describe treatment adherence to clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel in patients with acne vulgaris in Canadian routine clinical practice, as captured in a daily electronic diary using percentage of patients who achieve at least 80% treatment adherence at Week-4, Week-8, Week-12, and Week-20 from treatment initiation.
Treatment Effectiveness as assessed by mean change from baseline in Investigator Global Assessment (IGA) score | Baseline, Week-12, and Week-20
  To describe the effectiveness of clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel in patients with acne vulgaris in Canadian routine clinical practice, as assessed by mean change in IGA score at Week-12 and Week-20 from baseline. The IGA is a 5-point scale (0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe), with higher scores indicating worse acne severity.
Treatment Effectiveness as assessed by mean Investigator Global Assessment (IGA) score | Baseline, Week-12, and Week-20
  To describe the effectiveness of clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel in patients with acne vulgaris in Canadian routine clinical practice, as assessed by mean IGA score at baseline, Week-12, and Week-20. The IGA is a 5-point scale (0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe), with higher scores indicating worse acne severity.
Treatment Effectiveness as assessed by percentage of patients achieving at least a 1-grade improvement in Investigator Global Assessment (IGA) score | Baseline, Week-12, and Week-20
  To describe the effectiveness of clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel in patients with acne vulgaris in Canadian routine clinical practice, as assessed by the percentage of patients who have achieved at least a 1-grade improvement at Week-12 and Week-20 from baseline. The IGA is a 5-point scale (0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe), with higher scores indicating worse acne severity.
Treatment Effectiveness as assessed by number and percentage of patients achieving a score of 0 to 1 in Investigator Global Assessment (IGA) score | Week-12, and Week-20
  To describe the effectiveness of clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel in patients with acne vulgaris in Canadian routine clinical practice, as assessed by number and percentage of patients who achieve IGA = 0 to 1 at Week-12 and Week-20. The IGA is a 5-point scale (0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe), with higher scores indicating worse acne severity.
Safety and Tolerability | From baseline to Week-20
  To describe the safety and tolerability of clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel in patients with acne vulgaris in Canadian routine clinical practice, with number and percentage of adverse events (AEs) and serious AEs (SAEs) reported over 20 weeks, and number and percentage of patients who discontinued due to an AE or SAE at Week-20.
Health State Utility as assessed by Health Utility Index 2 (HUI2) | Baseline, Week-12, and Week-20
  To describe the health state utility scores in patients with acne vulgaris treated with clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel in Canadian routine clinical practice, as per percentage change in Health Utility Index 2 (HUI2) score at Week-12 and Week-20 from baseline, and mean HUI2 score at baseline, Week-12, and Week-20.

OTHER OUTCOMES:
Utilization Patterns of Cleanser, Moisturizer, and Sun Protectant | From Baseline to Week 20
  To describe the utilization patterns of cleanser, moisturizer, and sun protectant in patients with acne vulgaris treated with clindamycin phosphate 1.2% / adapalene 0.15% / benzoyl peroxide 3.1% gel in Canadian routine clinical practice, as captured in a daily electronic diary.

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Gaudet, Study Director — Bausch Health, Canada Inc.
Locations (18):
- Canada (18):
  - CHARM Site 001, Edmonton, Alberta
  - CHARM Site 017, Surrey, British Columbia
  - CHARM Site 012, Vancouver, British Columbia
  - CHARM Site 003, Winnipeg, Manitoba
  - CHARM Site 021, Hamilton, Ontario
  - CHARM Site 010, Markham, Ontario
  - CHARM Site 013, Newmarket, Ontario
  - CHARM Site 022, North York, Ontario
  - CHARM Site 015, Ottawa, Ontario
  - CHARM Site 011, Richmond Hill, Ontario
  - CHARM Site 016, Toronto, Ontario
  - CHARM Site 005, Toronto, Ontario
  - CHARM Site 014, Toronto, Ontario
  - CHARM Site 002, Toronto, Ontario
  - CHARM Site 019, Windsor, Ontario
  - CHARM Site 008, Montreal, Quebec
  - CHARM Site 006, Pointe-Claire, Quebec
  - CHARM Site 018, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided